CLINICAL TRIAL: NCT02024659
Title: Effects and Safety of Budesonide Inhalation Suspension Via Transnasal Nebulization in Eosinophilic Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Effects and Safety of Budesonide Inhalation Suspension Via Transnasal Nebulization in Nasal Polyps
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Luo Zhang, Director, Beijing Institute of Otolaryngology., Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TongRen-BJO
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Nasal Polyps
Keywords: nasal polyps; remodeling; inflammatory cells; budesonide
MeSH Terms: conditions — Nasal Polyps | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- budesonide (Experimental)
  Interventions: Drug: budesonide
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: budesonide — Patients receive 1mg/2ml budesonide twice daily via transnasal nebulization for 14 days.
  Arms: budesonide
Other: placebo — patients receive placebo (saline solution) 2ml twice daily for 14 days.
  Arms: placebo

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial enrolled subjects with eosinophilic CRSwNP. Subjects were randomized to receive either budesonide inhalation suspension or placebo for 14 days. Visual analogue scales (VAS）of nasal symptoms, endoscopic polyp scores and morning serum cortical levels were assessed pre- and post-treatment. Polyp samples were evaluated for inflammatory cytokines, matrix metalloproteinases (MMPs) and tissue inhibitors of metalloproteinases (TIMPs) by immunoassay; collagen by histochemistry; and frequencies of different inflammatory T cell infiltration by flow cytometry. this study is undertaken to evaluate the efficacy of short-term prescription of budesonide inhalation suspension via transnasal nebulization by clinical and immunologic assessments. As outcome parameters for remodeling, differences in the expression of collagen and albumin were investigated before and after budesonide treatment. Meanwhile, TGF-β, MMPs and TIMPs expression differences in nasal polyps were investigated to explore underlying mechanisms of tissue reconstitution.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic rhinosinusitis was made on the basis of symptoms of rhinosinusitis for at least 12 weeks, confirmed by abnormalities in all sinuses on computed tomography scan.
* Bilateral nasal polyps were present.
* CRSwNP was defined as eosinophilic when percent of tissue eosinophils exceeded 10% of total infiltrating cells.
* All patients had taken no steroids or antibiotics for at least 4 weeks before sample collection.

Exclusion Criteria:

* cystic fibrosis
* pregnancy
* serious or unstable concurrent disease
* psychological disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
reduction of nasal polyp size | from baseline to two weeks
  endoscopic polyp scores are assessed pre- and post-treatment.
patients' assessment of symptoms improvement | from baseline to two weeks
  Four major symptoms, including nasal obstruction, discharge, loss of smell, headache/ facial pain, and TNSS were assessed by the patient pre- and post-treatment

SECONDARY OUTCOMES:
immunologic effect of budesonide transnasal nebulization in CRSwNP | from baseline to 2 weeks
  Polyp samples were evaluated for inflammatory cytokines, mediators and cellular infiltration pre- and post-treatment.
remodeling effect of budesonide transnasal nebulization in CRSwNP | from baseline to 2 weeks
  Albumin, collagen,TGF-beta, matrix metalloproteinases (MMPs) and tissue inhibitors of metalloproteinases (TIMPs) were measured in tissue homogenate at baseline and after 2-week treatment

OTHER OUTCOMES:
safety of budesonide via transnasal nebulization in nasal polyps | from baseline to 2 weeks
  Morning corticol level is measured pre- and post-treatment. The incidence and severity of adverse events are recorded during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, MD, Principal Investigator — Beijing Institute of Otolaryngology
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China